CLINICAL TRIAL: NCT03010059
Title: An Open-label, Randomized, 3-way Crossover Study in Healthy Adult Subjects to Assess the Relative Bioavailability of a Single Dose of JNJ-64041575 Administered as 2 Different New Concept Formulations (Oral Suspension and Tablet) Compared to Their Respective Current Formulations, and to Assess the Effect of Food on the Pharmacokinetics of the 2 New Concept Formulations
Brief Title: A Study to Assess the Relative Bioavailability of JNJ64041575 Administered as 2 Different New Concept Formulations (Oral Suspension and Tablet) Compared to Their Respective Current Formulations, and to Assess the Effect of Food on the Pharmacokinetics of the 2 New Concept Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108251; 2016-004018-86 (EudraCT Number); 64041575RSV1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-01-03; First posted 2017-01-04 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Panel 1: Treatment ABC (Experimental): Participants will receive 240 milligram (mg) JNJ-64041575 as 6.0 milliliter (mL) of a 40-milligram per milliliter (mg/mL) current oral suspension formulation (reference 1) under fasted conditions (Treatment A) in period 1, then 4.0 mL of a 60-mg/mL new concept oral suspension formulation (test 1) under fasted conditions (Treatment B) in period 2 followed by 4.0 mL of a 60-mg/mL new concept oral suspension formulation (test 2) under fed conditions (Treatment C) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral suspension formulation)
- Panel 1: Treatment BCA (Experimental): Participants will receive Treatment B (test 1) in period 1, then Treatment C (test 2) in period 2 followed by Treatment A (reference 1) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral suspension formulation)
- Panel 1: Treatment CAB (Experimental): Participants will receive Treatment C (test 2) in period 1, then Treatment A (reference 1) in period 2 followed by Treatment B (test 1) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral suspension formulation)
- Panel 1: Treatment ACB (Experimental): Participants will receive Treatment A (reference 1) in period 1, then Treatment C (test 2) in period 2 followed by Treatment B (test 1) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral suspension formulation)
- Panel 1: Treatment BAC (Experimental): Participants will receive Treatment B (test 1) in period 1, then Treatment A (reference 1) in period 2 followed by Treatment C (test 2) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral suspension formulation)
- Panel 1: Treatment CBA (Experimental): Participants will receive Treatment C (test 2) in period 1, then Treatment B (test 1) in period 2 followed by Treatment A (reference 1) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral suspension formulation)
- Panel 2: Treatment DEF (Experimental): Participants will receive JNJ-64041575 as 1 tablet of the 250-mg current oral tablet formulation (reference 2) under fasted conditions (Treatment D) in period 1, then 1 tablet of the 250-mg new concept oral tablet formulation (test 3) under fasted conditions (Treatment E) in period 2 followed by 1 tablet of the 250-mg new concept oral tablet formulation (test 4) under fed conditions (Treatment F) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral tablet formulation )
- Panel 2: Treatment EFD (Experimental): Participants will receive Treatment E (test 3) in period 1, then Treatment F (test 4) in period 2 followed by Treatment D (reference 2) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral tablet formulation )
- Panel 2: Treatment FDE (Experimental): Participants will receive Treatment F (test 4) in period 1, then Treatment D (reference 2) in period 2 followed by Treatment E (test 3) then in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral tablet formulation )
- Panel 2: Treatment DFE (Experimental): Participants will receive Treatment D (reference 2) in period 1, then Treatment F (test 4) in period 2 followed by Treatment E (test 3) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral tablet formulation )
- Panel 2: Treatment EDF (Experimental): Participants will receive Treatment E (test 3) in period 1, then Treatment D (reference 2) in period 2 followed by Treatment F (test 4) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral tablet formulation )
- Panel 2: Treatment FED (Experimental): Participants will receive Treatment F (test 4) in period 1, then Treatment E (test 3) in period 2 followed by Treatment D (reference 2) in period 3 on Day 1. There will be a washout period of at least 14 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-64041575 (oral tablet formulation )

INTERVENTIONS:
Drug: JNJ-64041575 (oral suspension formulation) — Participants will receive 240 mg JNJ-64041575 under fasted and fed conditions in Panel 1 as current/new concept oral suspension formulation.
  Other Names: ALS-008176
  Arms: Panel 1: Treatment ABC; Panel 1: Treatment ACB; Panel 1: Treatment BAC; Panel 1: Treatment BCA; Panel 1: Treatment CAB; Panel 1: Treatment CBA
Drug: JNJ-64041575 (oral tablet formulation ) — Participants will receive 250 mg JNJ-64041575 under fasted and fed conditions in Panel 2 as current/new concept oral tablet formulation.
  Other Names: ALS-008176
  Arms: Panel 2: Treatment DEF; Panel 2: Treatment DFE; Panel 2: Treatment EDF; Panel 2: Treatment EFD; Panel 2: Treatment FDE; Panel 2: Treatment FED

SUMMARY:
The purpose of this study is to assess the rate and extent of absorption of JNJ-64041575 by measuring ALS-008112 plasma concentrations following administration of a single oral dose of JNJ-64041575 given as 2 new concept formulations (oral suspension and tablet) compared to their respective current formulations under fasted conditions and to assess the effect of food on the pharmacokinetics of the 2 new concept formulations under fed condition in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI; weight in kg divided by the square of height in meters) between 18.0 and 30.0 kilogram per square meter kg/m^2, extremes included, and a body weight not less than 50.0 kg, extremes included
* Participant must have a normal 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function at screening, including: a) normal sinus rhythm (heart rate between 45 and 100 beats per minute [bpm], extremes included); b) QT corrected according to Fridericia's formula (QTcF) interval less than or equal to (<=)430 milliseconds (ms) for male participants and <=450 ms for female participants; c) QRS interval <=110 ms; d) PR interval <=200 ms; e) ECG morphology consistent with healthy cardiac conduction and function. Any evidence of heart block, or of left or right bundle branch block is exclusionary
* Participants must have normal values for alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (less than or equal (<=)1.0×upper limit of laboratory normal range [ULN])
* Contraceptive use by female participants should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies. Before randomization, a woman must be either: a) Not of childbearing potential defined as: 1) Postmenopausal: A postmenopausal state is defined as greater than (>)45 years and no menses for 12 consecutive months without an alternative medical cause and a serum follicle stimulating hormone (FSH) level in the postmenopausal range (>40 International units per liter [IU/L] or milli-international units per milliliter [mIU/mL]), OR; 2) Permanently sterile: Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures (without reversal operation), and bilateral oophorectomy b) Of childbearing potential and, if heterosexually active, 1) Practicing a highly effective method of contraception (failure rate of less than (<)1percent (%) per year when used consistently and correctly) 2) Agrees to remain on a highly effective method throughout the study and for at least 44 days after the last dose of study drug
* A female participant, except if postmenopausal, must have a negative serum beta human chorionic gonadotropin (beta- hCG) pregnancy test at screening, and a negative urine pregnancy test on Day 1 in each treatment period
* Participant must be able to taste and smell normally, to their own opinion. Participants who have an impaired sense of taste and/or smell due to any conditions such as allergic rhinitis, common cold, or sinusitis are not eligible to take part in the study

Exclusion Criteria:

* Participant has a mouth pathology including, but not limited to, pain, ulcer, edema, mucosal erosion, gingivitis and/or (dental) abscesses, or receives treatment for oral pathologies (eg, antifungals or antibiotics) or oral treatment for any disease
* Participant with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs
* Participant is hepatitis B surface antigen (HBsAg) positive or hepatitis C virus (HCV) antibody positive with HCV RNA positive, or has another clinically active liver disease at screening
* Participant has a history of human immunodeficiency virus type 1 (HIV-1) or HIV 2 antibody positive, or tests positive for HIV-1 or -2 at screening
* Participant has previously been dosed with JNJ-64041575 in more than 3 single-dose studies with JNJ-64041575 or has previously been dosed with JNJ-64041575 in a multiple-dose study with JNJ-64041575
* Participants with 1 or more of the following laboratory abnormalities at screening as defined by the Division of Microbiology and Infectious Diseases (DMID) Adult Toxicity Table a) Serum creatinine grade 1 or greater (greater [>]1.0* upper limit of laboratory normal range [ULN]) b) Hemoglobin grade 1 or greater (<=10.5 gram per decilitre [g/dL]) c) Platelet count grade 1 or greater (<=99.999/millimeter [mm]^3) d) Reticulocyte count (absolute) below the lower limit of laboratory normal range (LLN) e) Absolute neutrophil count grade 1 or greater (<=1,500/mm^3) f) Total bilirubin grade 1 or greater (>1.0*ULN) g) Any other toxicity grade 2 or above, except for grade 2 elevations of low density lipoprotein (LDL) cholesterol and/or cholesterol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ALS-008112 (JNJ-63549109) | Up to Day 8
  Cmax is the maximum observed plasma concentration.
Area Under Plasma Concentration Curve from time zero to the last quantifiable (AUC [0-last]) of ALS-008112 (JNJ-63549109) | Up to Day 8
  Area under the plasma concentration time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non BQL]) concentration, calculated by linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of ALS-008112 (JNJ-63549109) | Up to Day 8
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/ lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.

SECONDARY OUTCOMES:
Time to Reach Maximum Concentration (Tmax) ALS-008112 (JNJ-63549109) | Up to Day 8
  Tmax is defined as actual sampling time to reach maximum observed plasma concentration.
Apparent Terminal Elimination Rate Constant (lambda z) of ALS-008112 (JNJ-63549109) | Up to Day 8
  Apparent terminal elimination rate constant, determined by linear regression using the terminal log linear phase of the log transformed concentration versus time curve.
Apparent Terminal Elimination Half-life (t1/2term) of ALS-008112 (JNJ-63549109) | Up to Day 8
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration time curve and calculated as 0.693/apparent terminal elimination rate constant (lambda[z]).
Maximum Observed Plasma Concentration (Cmax) of ALS-008144 (JNJ-64167896) | Up to Day 8
  Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Concentration (Tmax) of ALS-008144 (JNJ-64167896) | Up to Day 8
  Tmax defined as the actual sampling time to reach the maximum observed plasma concentration.
Area Under Plasma Concentration Curve from time zero to the last quantifiable (AUC [0-last]) of ALS-008144 (JNJ-64167896) | Up to Day 8
  AUC (0-last) defined as area under the plasma concentration time curve (AUC) from time 0 to the time of the last measurable (non below quantification limit [non-BQL]) concentration, calculated by linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of ALS-008144 (JNJ-64167896) | Up to Day 8
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time calculated as the sum of AUC (0-last) and C (0-last)/ lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(0-last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Apparent Terminal Elimination Rate Constant (lambda z) of ALS-008144 (JNJ-64167896) | Up to Day 8
  Apparent terminal elimination rate constant, determined by linear regression using the terminal log linear phase of the log transformed concentration versus time curve.
Apparent Terminal Elimination Half-life (t1/2term) of ALS-008144 (JNJ-64167896) | Up to Day 8
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration time curve and calculated as 0.693/apparent terminal elimination rate constant (lambda[z]).
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Screening (28 days ) to Follow up Phase (10 to 14 days after last dose)
  Safety and Tolerability
Taste of JNJ-64041575 following administration of different oral suspension formulations under fed and fasted conditions in healthy adult participants in Panel 1 (taste questionnaire) | Day 1
  Participants will complete a taste questionnaire within 5 to 15 minutes after study drug intake in each treatment period. For the taste questionnaire, a dichotomization will be made for the overall question, categorizing 'bad' and 'almost acceptable' versus 'acceptable' and 'good'.
Taste and Swallowability of JNJ-64041575 following administration of different oral tablet formulations under fed and fasted conditions in healthy adult participants in Panel 2 (taste and swallowability questionnaire) | Day 1
  A taste and swallowability questionnaire will be completed by the participant within 5 to 15 minutes after each study drug intake in each treatment period, to compare the taste and swallowability (tablets only) of JNJ-64041575 following administration of different oral formulations under fed and fasted conditions. For the taste questionnaire, a dichotomization will be made for the overall question, categorizing 'bad' and 'almost acceptable' versus 'acceptable' and 'good'. For the swallowability, a dichotomization will be made of 'slightly difficult' or worse versus 'neither difficult nor easy' or better. The results of the questionnaire will be transcribed into the e-Source by a member of the study-site personnel.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium